CLINICAL TRIAL: NCT03887065
Title: Magnetic Resonance Imaging 12 Day Study for Multiple Sclerosis/Clinically Isolated Syndrome Trial of JM-4 Novel Human Peptide
Brief Title: Magnetic Resonance Imaging Study of JM-4 in Multiple Sclerosis/Clinically Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cook, Stuart, MD (Other)
Responsible Party: Principal Investigator, Stuart Cook, MD, Professor, Cook, Stuart, MD
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JM-4-001
Record Dates: First submitted 2019-03-10; First posted 2019-03-22 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Starting dose (Experimental): Three to five patients will receive a daily dose of 1 mg/kg JM-4 (in normal saline) delivered via intravenous infusion for no more than 30 minutes for up to 7 consecutive days.
  Interventions: Drug: JM-4
- Intermediate dose of JM-4 (Experimental): Three to five patients will receive a daily dose of 4 mg/kg of JM-4 (in normal saline) via intravenous infusion for no more than 30 minutes for up to 7 consecutive days.
  Interventions: Drug: JM-4
- High dose of JM-4 (Experimental): Three to five patients will receive a daily dose of 9 mg/kg of JM-4 (in normal saline) via intravenous infusion for no more than 30 minutes for up to 7 consecutive days.
  Interventions: Drug: JM-4

INTERVENTIONS:
Drug: JM-4 — Novel small human peptide derived from erythropoietin

SUMMARY:
This is a Phase 0/1 study of MS patients to determine the safety and potential efficacy of a novel, small human peptide designated as JM-4. The study will involve treatment for 5-7 days with JM-4 to determine the effects of Gadolinium(+) lesion number and volume in the brains of patients.

DETAILED DESCRIPTION:
This study is the first study of JM-4 in patients with Multiple Sclerosis and is intended to show safety and potential efficacy in changing the size and/or number of GAD(+) lesions in the brain. The initial dose level of 1 mg/kg/ will establish safety of JM-4 treatment after 5-7 days of treatment via intravenous infusion over 30 minutes daily in3-5 patients with Multiple Sclerosis. MRI examinations will be conducted prior to treatment with JM-4 and 8 days after the initiation of treatment for the purpose of quantitating GAD(+) brain lesions. Once initial safety is established, the next group of 3-5 patients will receive 4 mg/kg/ of JM-4 daily for 5-7 days via 30 minute intravenous infusions, with MRI scans conducted prior to treatment and 8 days after the initial dose of JM-4. Once safety is established in this cohort of patients, a third group of patients may receive 9 mg/kg/ of JM-4 daily for 5-7 days via 30 minute infusions, with MRI scans conducted prior to the initial treatment and 8 days after the initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS (McDonald criteria) or CIS
* GAD(+) MRI brain lesion on screening exam, with or without clinical activity followed by a baseline MRI
* EDSS of 0-5.5 inclusive
* Weight of 40-115 kg
* Females must be post-menopausal or surgically sterilized or use a hormonal contraceptive, intra-uterine device or diaphragm with spermicide during the study
* Not be pregnant or breast feeding
* Males must be willing to use contraception during each day of the study
* Be willing to comply with study procedures and protocols for the duration of the study
* Voluntarily provide informed consent
* Be wiling and physically able to attend the study center as required for all study screening and procedures

Exclusion Criteria:

* Taking Tysabri, Gilenya, Tecfidera, Aubagio, Ocrevus or other immunosuppressive drugs within the prior 3 months
* Received Mitoxantrone or Lemtrada at any time
* Consumption of corticosteroids within the past 30 days
* Current or less than 5 years prior malignancy (excluding basal cell or squamous cell skin cancer)
* Serious systemic disorder which might, in the opinion of the investigators, interfere with safety, compliance, treatment or evaluation of efficacy. Conditions would include but not be limited to significant cardiac, liver, kidney, lung or cerebrovascular disease, HIV, serious infections, serous psychiatric disease or poorly controlled diabetes mellitus
* aversion, intolerance or allergy to repeated MRI with gadolinium administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-06-15 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events | From initial dose through 8 days after initiation of dosing
  To determine the incidence of adverse events and any abnormal laboratory values
Change in GAD(+) brain lesions measured via MRI scan | From initial dose through 8 days after initiation of dosing
  Measurement of the number and size of GAD(+) brain lesions from baseline to post-dosing 8 days after initiation of treatment

SECONDARY OUTCOMES:
Changes in the ability of patients to complete a timed 25-foot walk | From initial dosing through 8 days post-initiation of dosing
  To determine changes in timed 25 foot walk prior to treatment or 8 days after treatment
Treatment-induced changes in Expanded Disability Status Score in patients | Prior to initial dose through 8 days post-initial treatment
  Measurement of Expanded Disability Status scores in patients prior to treatment and after completion of treatment
Changes in neurological exam | Prior to initial dose through 8 days post-initial treatment
  Neurological examination of patients to check for optic nerve changes and vision changes

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Cook, MD, Principal Investigator — VA Medical Center

IPD SHARING:
Plan to Share IPD: No